CLINICAL TRIAL: NCT04528901
Title: Study of seroPREvalence Vis-à-vis SARS-CoV2 and Correlation With Clinical Forms of COVID-19 in Patients Followed in Pneumology in the Cluster Area of the Grand-Est Region (Strasbourg University Hospital)
Acronym: PRESAGE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7879
Record Dates: First submitted 2020-08-25; First posted 2020-08-27 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2020-09

CONDITIONS: Covid-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
seroPREvalence vis-à-vis SARS-CoV2 and correlation with clinical forms of COVID-19 in patients followed in Pulmonology in the cluster area of the Grand-Est region.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman from 18 years old and without upper age limit
* Patient followed in pulmonology at Strasbourg University Hospital
* Patient presenting at least one of the following pathologies:

  1. severe persistent asthma (200 patients)
  2. chest cancer that is active or has received treatment within a period of less than one year (300 patients)
  3. history of lung transplantation performed before the start of the epidemic (02/29/2020) (300 patients)
  4. idiopathic or other diffuse interstitial lung disease, sarcoidosis or vasculitis (70 patients)
  5. pulmonary arterial hypertension (PAH) (group 1 of the international classification) any cause or chronic thromboembolic PAH (group 4): (60 patients)
  6. Severe COPD in the respiratory failure stage (150 patients)
* Subject affiliated to a social health insurance protection scheme
* Subject able to understand the objectives of the research
* Subject having signed an informed consent

Exclusion Criteria:

* Inability to provide informed information about the subject (subject in an emergency situation, difficulty in understanding the subject, etc.)
* Subject under safeguard of justice
* Subject under guardianship or guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient followed in pulmonology at Strasbourg University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 1080 (Estimated)
Dates: Start 2020-09-04 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Determine and compare the seroprevalence for SARS-CoV2 among patients with respiratory pathologies monitored in Pneumology at the Strasbourg University Hospital, in the cluster zone of the Grand Est. | 15 months
  Carrying out a serological assay of specific antibodies to SARS-CoV-2

CONTACTS AND LOCATIONS:
Overall Officials: Céline MASCAUX, Principal Investigator — CHU de Strasbourg
Locations (1):
- Les Hôpitaux Universitaires de Strasbourg, Strasbourg, Bas-Rhin, France

IPD SHARING:
Plan to Share IPD: Undecided